CLINICAL TRIAL: NCT01363050
Title: A Phase 1, Open Label, Multiple Dose Study to Determine the Tolerability, Safety and Pharmacokinetics of Ketorolac Tromethamine by Intranasal Administration in Healthy Volunteers
Brief Title: Study to Determine the Tolerability, Safety and Pharmacokinetics of Ketorolac Tromethamine by Intranasal Administration in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Egalet Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROX 2005-03
Record Dates: First submitted 2011-05-27; First posted 2011-06-01 (Estimated); Results first posted 2013-05-03 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Ketorolac Tromethamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ketorolac tromethamine (Experimental)
  Interventions: Drug: Ketorolac tromethamine

INTERVENTIONS:
Drug: Ketorolac tromethamine — Subjects received intranasal ketorolac tromethamine (30 mg) three times daily (t.i.d.) for three days (seven doses in total). Doses were administered every eight hours.

SUMMARY:
This was a phase 1, open label, multiple dose study in healthy male and female volunteers. Subjects received intranasal ketorolac tromethamine (30 mg) three times daily (t.i.d.) for three days (seven doses in total). Doses were administered every eight hours.

The objective of this study in healthy volunteers was to determine the safety, tolerability, and pharmacokinetics of multiple doses of intranasal ketorolac tromethamine.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers, aged 18 to 60 years inclusive
* Female subjects of child bearing potential were to have a negative urine pregnancy test prior to entry into the study and must not have been breast feeding
* All female subjects of child bearing potential and all male subjects with female partners of child bearing potential must have consented to using a medically acceptable method of contraception (oral or implanted contraceptive hormones, condom or diaphragm with spermicidal agent, intrauterine device or surgical sterilisation) throughout the study period
* Subject had given signed informed consent
* Subject was within 20% of normal weight for his/her height and body build according to the table of "Desirable Weights for Men and Women" (Metropolitan Life Insurance Co. 1999)
* Subject's medical history was considered normal, with no clinically significant abnormalities
* Subject was considered to be in good health in the opinion of the Investigator, as determined by a pre-study physical examination with no clinically significant abnormalities, vital signs within normal ranges and an ECG with no clinically significant abnormalities
* Subject's pre-study clinical laboratory findings were within normal range or, if outside of the normal range, not deemed clinically significant in the opinion of the Investigator
* Subject had bilateral patent nasal airways at screening as assessed by the Investigator
* Body weight of at least 60 kg

Exclusion Criteria:

* Subject had a clinically significant illness in the four weeks prior to screening
* Use of prescribed medications in the three weeks prior to dosing or over-the-counter preparations for seven days prior to dosing, except paracetamol which was allowed up to 48 hours prior to dosing. Use of multivitamins and oral contraceptives were permitted
* Subject had a significant history of drug/solvent abuse, or a positive drugs of abuse test at screening
* Subjects with a history of alcohol abuse or those currently drinking more than 28 units per week (males) or 21 units per week (females)
* Current tobacco use or a history of smoking within the past five years
* Subject was, in the opinion of the Investigator, not suitable to participate in the study
* Subjects who had participated in any clinical study with an investigational drug/device within three months prior to the first day of dosing
* Subjects who had a positive result of HIV screen, Hepatitis B screen or Hepatitis C screen
* Subjects who had a serious adverse reaction or significant hypersensitivity to any drug
* Subjects having donated 500 mL or more of blood within the three months prior to screening
* Any history of co-existing nasal polyps, NSAID sensitivity and asthma
* Allergic reaction to aspirin or other NSAIDs
* Current upper respiratory tract infection or other respiratory tract condition that may have interfered with the absorption of the nasal spray or with the assessment of adverse events (AEs)
* Any suspicion of rhinitis medicamentosa (chronic daily use of topical decongestants)
* Use of a monoamine oxidase inhibitor (MAOI) in the 14 days prior to study entry
* Active peptic ulcer disease, gastrointestinal bleeding or perforation, or a history of peptic ulcer disease or gastrointestinal bleeding
* Anemia due to unexplained or known gastrointestinal bleeding
* History of asthma or any other chronic pulmonary disorder
* Renal impairment or a risk of renal failure due to volume depletion
* Known sensitivity to lidocaine hydrochloride

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2006-01; Primary Completion 2006-02 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cyril Clarke, BSc MB BS MFPM, Principal Investigator — Medeval Limited
Locations (1):
- Medeval Limited, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: January 9, 2006 - February 27, 2006; Clinical Unit
Pre-assignment Details: After subjects had given their informed consent, subjects were required to pass a screening visit within 3 weeks prior to study drug administration.
Groups:
- Ketorolac Tromethamine: Ketorolac tromethamine : Subjects received intranasal ketorolac tromethamine (30 mg) three times daily (t.i.d.) for three days (seven doses in total). Doses were administered every eight hours.
Period: Overall Study
Arm/Group | Ketorolac Tromethamine
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ketorolac Tromethamine
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Region of Enrollment [Number; unit: participants]
  United Kingdom | 15

OUTCOME MEASURES:

1. Primary Outcome: Cmax (the Maximum Observed Plasma Concentration)
Description: PK analysis by standard model independent methods was performed by a pharmacokineticist using WinNonlin Professional. Actual blood sampling times were converted to a time from dosing (elapsed time). Elapsed times were listed by subject for each treatment, together with the individual plasma concentrations of ketorolac.
Time Frame: Blood samples for determination of plasma concentration of ketorolac were taken immediately prior to each dose and every hour for 8 hours post-dose on Day 1 (morning doses)
Population: Two subjects were considered pharmacokinetic outliers and were excluded from the PK population.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Ketorolac Tromethamine: Ketorolac tromethamine (Day 1) : Subjects received intranasal ketorolac tromethamine (30 mg) three times daily (t.i.d.) for three days (seven doses in total). Doses were administered every eight hours.
Arm/Group | Ketorolac Tromethamine
Number analyzed (Participants) | 13
ng/mL | 1147.9 (186.0)

2. Primary Outcome: Tmax (the Time to Maximum Concentration)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Two subjects were considered pharmacokinetic outliers and were excluded from the PK population.
Measure: Median (Full Range); unit: hours
Arm/Group | Ketorolac Tromethamine
Number analyzed (Participants) | 13
hours | 1.000 [1.00 to 7.92]

3. Primary Outcome: AUC 0-8h (the Area Under the Plasma Concentration-time Curve From Time 0 to 8 Hours Post-dose)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Two subjects were considered pharmacokinetic outliers and were excluded from the PK population.
Measure: Mean (Standard Deviation); unit: ng*hours/mL
Groups:
- Ketorolac Tromethamine: Ketorolac tromethamine (Day 1): Subjects received intranasal ketorolac tromethamine (30 mg) three times daily (t.i.d.) for three days (seven doses in total). Doses were administered every eight hours.
Arm/Group | Ketorolac Tromethamine
Number analyzed (Participants) | 13
ng*hours/mL | 4713.8 (744.8)

4. Primary Outcome: Cmax,ss (the Maximum Observed Plasma Concentration at Steady State)
Description: as for outcome 1
Time Frame: Blood samples for determination of plasma concentration of ketorolac were taken immediately prior to each dose and every hour for 8 hours post-dose on Day 3 (morning doses)
Population: Two subjects were considered pharmacokinetic outliers and were excluded from the PK population.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Ketorolac Tromethamine: Ketorolac tromethamine (Day 3): Subjects received intranasal ketorolac tromethamine (30 mg) three times daily (t.i.d.) for three days (seven doses in total). Doses were administered every eight hours.
Arm/Group | Ketorolac Tromethamine
Number analyzed (Participants) | 13
ng/mL | 1382.6 (224.3)

5. Primary Outcome: Tmax,ss (the Time to Maximum Concentration at Steady State)
Description: as for outcome 1
Time Frame: as for outcome 4
Population: Two subjects were considered pharmacokinetic outliers and were excluded from the PK population.
Measure: Median (Full Range); unit: hours
Arm/Group | Ketorolac Tromethamine
Number analyzed (Participants) | 13
hours | 1.000 [1.00 to 3.00]

6. Primary Outcome: Cmin,ss (the Minimum Observed Plasma Concentration at Steady State)
Description: as for outcome 1
Time Frame: as for outcome 4
Population: Two subjects were considered pharmacokinetic outliers and were excluded from the PK population.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ketorolac Tromethamine
Number analyzed (Participants) | 13
ng/mL | 367.7 (67.7)

7. Primary Outcome: Tmin,ss (the Time to Minimum Concentration at Steady State)
Description: as for outcome 1
Time Frame: as for outcome 4
Population: Two subjects were considered pharmacokinetic outliers and were excluded from the PK population.
Measure: Median (Full Range); unit: hours
Arm/Group | Ketorolac Tromethamine
Number analyzed (Participants) | 13
hours | 0.000 [0.00 to 8.00]

8. Primary Outcome: AUCτ (the Area Under the Plasma Concentration-time Curve Over the Dosing Interval at Steady-state)
Description: as for outcome 1
Time Frame: as for outcome 4
Population: Two subjects were considered pharmacokinetic outliers and were excluded from the PK population.
Measure: Mean (Standard Deviation); unit: ng*hours/mL
Arm/Group | Ketorolac Tromethamine
Number analyzed (Participants) | 13
ng*hours/mL | 6379.2 (1031.0)

9. Primary Outcome: MRT (the Mean Residence Time
Description: as for outcome 1
Time Frame: as for outcome 4
Population: Two subjects were considered pharmacokinetic outliers and were excluded from the PK population.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ketorolac Tromethamine
Number analyzed (Participants) | 13
hours | 3.368 (0.056)

ADVERSE EVENTS:
Time Frame: 1 month and 3 weeks
Arm/Group | Ketorolac Tromethamine
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 14/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketorolac Tromethamine (N=15)
Lacrimation increased (Eye disorders) | 2 (4)
Lip dry (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Catheter site haematoma (General disorders) | 1 (1)
Feeling cold (General disorders) | 1 (1)
Rhinitis (Infections and infestations) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (4)
Paraesthesia (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 4 (10)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Orthostatic hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No